CLINICAL TRIAL: NCT01805557
Title: Phase II Randomized Study With R-DHAP +/- Bortezomib as Induction Therapy in Relapsed/Refractory Diffuse Large B-cell Lymphoma (DLBCL) Patients Eligible to Transplantation. BR-DHAP Versus R-DHAP.
Acronym: FIL_VERAL12
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Fondazione Italiana Linfomi - ETS (Other)
Collaborators: Janssen Pharmaceutica (Industry); Janssen-Cilag Ltd. (Industry); Centro di Riferimento per l'Epidemiologia e la Prev. Oncologica Piemonte (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FIL_VERAL12
Record Dates: First submitted 2013-03-05; First posted 2013-03-06 (Estimated); Last update posted 2022-06-08 (Actual); Status verified 2022-06

CONDITIONS: Diffuse Large B-cell Lymphoma Refractory; Diffuse Large B-cell Lymphoma Recurrent
Keywords: Diffuse Large B-cell Lymphoma (DLBCL); Bortezomib
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- R-DHAP (Active Comparator): R-DHAP x 2, restaging, mobilization and harvest of peripheral stem cell + R-DHAP x 2, restaging with PET evaluation
  Interventions: Drug: R-DHAP
- BR-DHAP (Experimental): Bortezomib + R-DHAP x 2, restaging, mobilization and harvest of peripheral stem cell + Bortezomib + R-DHAP x 2, restaging with PET evaluation
  Interventions: Drug: R-DHAP; Drug: BR-DHAP

INTERVENTIONS:
Drug: R-DHAP — * Rituximab 375 mg/sqm iv day 0 or 1
  * Cisplatin 100 mg/sqm iv day 1 in 6-hours infusion
  * Cytarabine 2000 mg/sqm in 3-hours infusion iv day 2 and day 3
  * Dexamethasone 40 mg day 1-4
  * Pegfilgrastim 6 mg sc monodose 24 hours after the end of chemotherapy or G-CSF from day 5 till stem cell harvest during mobilization's course (II o III cycle R-DHAP)
  * Rituximab 375 mg/sqm iv 24 hours before apheresis as purging in vivo during second courses of therapy
Drug: BR-DHAP — * Rituximab 375 mg/sqm iv day 0 or 1
  * Bortezomib SC 1.5 mg/sqm day 1, day 4
  * Cisplatin 100 mg/sqm iv day 1 in 6-hours infusion
  * Cytarabine 2000 mg/sqm in 3-hours infusion iv day 2 and day 3
  * Dexamethasone 40 mg day 1-4
  * Pegfilgrastim 6 mg sc monodose 24 hours after the end of chemotherapy or G-CSF from day 5 till stem cell harvest during mobilization's course (II o III cycle R-DHAP)
  * Rituximab 375 mg/sqm iv 24 hours before apheresis as purging in vivo during second courses of therapy Chemotherapy R-DHAP and BR-DHAP will be repeated every 28 days.
  Arms: BR-DHAP

SUMMARY:
The probability to achieve CR with R-chemotherapy in patients failing a rituximab containing first line regimen is quite low, in particular in cases with non GCB profile. The bioCORAL trial suggest that ABC subset have a dismal outcome whichever the induction treatment. Thus it can be argued the addition of new molecule to the RDHAP regimen could be of value. Bortezomib appears the best candidate in this setting as ABC subtypes constitutively express NFkb, which is the target of bortezomib itself. Data from the literature suggest an encouraging activity of R-chemo+ bortezomib in non GCB-derived DLBCL, although in small series. Thus, the addition of bortezomib is here justified by the need to circumvent constitutional resistance to chemotherapy. Published experience of the association between bortezomib and cytarabine are also encouraging with acceptable cumulative toxicity.

DETAILED DESCRIPTION:
This is a prospective, multicenter, two-arm randomized phase II screening trial34 in young patients (18-65 years) affected by relapsed/refractory Diffuse Large B-cell Lymphoma (DLBCL) at diagnosis, eligible to high-dose therapy.

Aim of the study is to to assess whether the addition of Bortezomib to R-DHAP is more promising than standard R-DHAP, as induction therapy before high dose chemotherapy with ASCT with respect to response and safety. Patients will be randomized at first relapse between: a) the standard salvage therapy Rituximab in association to DHAP every 28 days (R-DHAP) for 4 cycles and b) Bortezomib in association to the same regimen (BR-DHAP). In both arms the induction therapy is followed by autologous stem cell transplantation or, if indicated, by allogeneic stem cell transplant.

A patient is considered evaluable if it is possible to assess response by PET after 4 cycle or, if a patient withdraws from the study for PD, before completion of study treatment.

After providing written informed consent, patients will be evaluated for eligibility during a 21-day screening period. If they continue to meet eligibility criteria, they will be randomized to receive the first dose of BR-DHAP or R-DHAP .

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-65
2. Relapsed/refractory disease after receiving one line of standard chemoimmunotherapy (R-CHOP, GA-CHOP, R-CHOP like)
3. Diffuse Large B-cell Lymphoma at relapse. Patient has to be re-biopsied prior to study entry. If this is harmful for the patient, the patient can be enrolled if archivial tumor sample and block from first diagnosis are available.
4. No prior Bortezomib therapy
5. Measurable and/or evaluable disease
6. Any Ann Arbor stage and IPI group at relapse
7. Performance status < 2 according to ECOG scale unless due to lymphoma
8. No Central Nervous System (CNS) disease (meningeal and/or brain involvement by lymphoma)
9. Adequate hematological counts: ANC > 1.5 x 109/L, Hgb > 9 g/dl (transfusion independent), Platelet count > 75 x 109/L (transfusion independent), with the exception of cytopenia due to lymphoma bone marrow involvement
10. HIV negativity, HCV negativity, HBV negativity or patients with HBcAb +, HBsAg -, HBs Ab+/- with HBV-DNA negativity (in these patients Lamivudine prophylaxis is mandatory)
11. Normal liver function (ALP, AST, ALT, GGT, conjugated bilirubin total < 2 x ULN) if not related to lymphoma
12. Normal kidney function (creatinine clearance > 45 ml/min)
13. Cardiac ejection fraction > 50% (MUGA scan or echocardiography)
14. Normal lung function
15. Absence of active opportunistic infections
16. Non peripheral neuropathy or active neurological non neoplastic disease of CNS
17. Non major surgical intervention prior 3 months to randomization if not due to lymphoma and/or no other disease life-threatening that can compromise chemotherapy treatment
18. Disease free of prior malignancies other than lymphoma for > 3 years with exception of currently treated squamous cell and basal cell carcinoma of the skin or carcinoma in situ of the cervix or breast
19. Life expectancy > 6 months
20. No psychiatric illness that precludes understanding concepts of the trial or signing informed consent
21. Written informed consent
22. Women must be:

    * postmenopausal for at least 1 year (must not have had a natural menses for at least 12 months)
    * surgically sterile (have had a hysterectomy or bilateral oophorectomy, tubal ligation, or otherwise be incapable of pregnancy),
    * abstinent (at the discretion of the investigator/per local regulations), or
    * if sexually active, be practicing a highly effective method of birth control (eg, prescription oral contraceptives, contraceptive injections, contraceptive patch, intrauterine device, double-barrier method (eg, condoms, diaphragm, or cervical cap, with spermicidal foam, cream, or gel, male partner sterilization) as local regulations permit, before entry, and must agree to continue to use the same method of contraception throughout the study. They must also be prepared to continue birth control measures for at least 12 months after terminating treatment.
23. Women of childbearing potential must have a negative serum or urine beta-human chorionic gonadotropin (beta-hCG) pregnancy test at screening
24. Men must agree to use an acceptable method of contraception (for themselves or female partners as listed above) for the duration of the study. Men must agree to use a double barrier method of birth control and to not donate sperm during the study and for 3 months after receiving the last dose of study drug.

Exclusion criteria:

1. Diagnosis of Lymphoblastic Lymphoma, Burkitt Lymphoma, Non Hodgkin Lymphoma CD20 negative, Mantle Cell Lymphoma, Follicular Lymphoma g I-II-IIIa-IIIb, Primary Mediastinal Lymphoma
2. Age > 65 years
3. Patients ineligible to high-dose chemotherapy
4. Performance status > 2 according to ECOG scale if not due to lymphoma
5. Patient has known or suspected hypersensitivity or intolerance to Rituximab
6. Patient has received an experimental drug or used an experimental medical device within 4 weeks before the planned start of treatment. Concurrent participation in non-treatment studies is allowed, if it will not interfere with participation in this study.
7. CNS disease (meningeal and/or brain involvement by lymphoma)
8. History of clinically relevant liver or renal insufficiency; significant cardiac, vascular, pulmonary, gastrointestinal, endocrine, neurologic, rheumatologic, hematologic, psychiatric, or metabolic disturbances
9. Uncontrolled diabetes (if receiving antidiabetic agents, subjects must be on a stable dose for at least 3 months before first dose of study drug
10. Uncontrolled or severe cardiovascular disease including myocardial infarction within six months of enrollment, New York Heart Association (NYHA) Class III or IV heart failure, uncontrolled angina, clinically significant pericardial disease, or cardiac amyloidosis
11. Cardiac ejection fraction < 50% (MUGA scan or echocardiography)
12. Creatinine clearance < 45 ml/min
13. Presence of major neurological disorders
14. HIV positivity, HCV positivity, HBV positivity with the exception of patients with HBcAb +, HbsAg -, HBs Ab+/- with HBV-DNA negative
15. Active opportunistic infection
16. Major surgical intervention prior 3 months to randomization if not due to lymphoma and/or other disease life-threatening that can compromise chemotherapy treatment
17. Prior malignancies other than lymphoma in the last 3 years with exception of currently treated squamous cell and basal cell carcinoma of the skin or carcinoma in situ of the cervix or breast
18. Life expectancy < 6 months
19. Any other coexisting medical or psychological condition that would preclude participation in the study or compromise ability to give informed consent.
20. If female, the patient is pregnant or breast-feeding.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2013-02-04 (Actual); Primary Completion 2019-03-12 (Actual); Study Completion 2020-11-20 (Actual)

PRIMARY OUTCOMES:
Complete Response (CR) Rate | At the end of the induction phase (6 months)
  Proportion of CR according to the Cheson 2007 response criteria, evaluated by PET scan

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | At the end of the induction phase (6 months)
  ORR at the end of the induction treatment is defined as Complete Response (CR) or Partial Response according to the Cheson 2007 response criteria, evaluated by PET scan
Overall Survival (OS) | 36 months
  OS will be defined as the time between the date of randomization and the date of death from any cause
Number of Patients With Treatment-Related Adverse Events (AEs)/Serious Adverse Events (SAEs) as a Measure of Safety | 12 months
  Incidence of grade 3 or higher Toxicity measured by CTCAE v.4 during therapy
Mobilizing potential | 6 months
  Amount of CD34+ stem cell collected/Kg
Number of Patients completing ASCT | 12 months
  Proportion of randomized patients successfully completing ASCT

CONTACTS AND LOCATIONS:
Overall Officials: Umberto Vitolo, MD, Study Director — SC Ematologia 2-AO Città della Salute e della Sienza-Molinette
Locations (24):
- Italy (24):
  - Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori-Ematologia, Meldola, Forlì-Cesena
  - Clinica Humanitas, Rozzano, Milano
  - ASST Grande Ospedale Metropolitano Niguarda - SC Ematologia, Milan, MI
  - CRO Aviano, Aviano, Pordenone
  - ASST Valle Olona, Gallarate, Varese
  - A.O. SS. Antonio e Biagio e C. Arrigo, Alessandria
  - Clinica di ematologia AOU Umberto I Ospedali Riuniti, Ancona
  - ASST Spedali Civili di Brescia - Ematologia, Brescia
  - Ospedale Businco - SC Ematologia e CTMO, Cagliari
  - Ematologia 1 Ospedale S. Martino, Genova
  - SC Ematologia - Trapianto di midollo osseo Fond. IRCCS Istituto Nazionale Tumori, Milan
  - SCDU Ematologia - Università del Piemonte Orientale, Novara
  - Ospedale S. Antonio, Padua
  - U.O. Complessa di Ematologia Ospedale di Parma, Parma
  - Ospedale Civile Guglielmo da Saliceto, Piacenza
  - Osp. S. Maria delle Croci, Ravenna
  - Grande Ospedale Metropolitano Bianchi Melacrino Morelli - Ematologia, Reggio Calabria
  - AO Arcispedale S.Maria Nuova Ematologia, Reggio Emilia
  - Osp. degli Infermi Divisione di Oncologia, Rimini
  - A.O. Universitaria S. Andrea, Roma
  - SC Oncoematologia con autotrapianto AO Santa Maria, Terni
  - AOU Citta della Salute e della Scienza di Torino - Ematologia Universitaria, Torino
  - AOU Citta della Salute e della Scienza di Torino-SC Ematologia, Torino
  - Azienda Ospedaliero - Universitaria di Udine, Udine

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-11-11): https://cdn.clinicaltrials.gov/large-docs/57/NCT01805557/Prot_SAP_000.pdf